CLINICAL TRIAL: NCT06697327
Title: Daunorubicin Plus Cytarabine 3+5 Regimen Combined With Venetoclax in de Novo Patients With Acute Myeloid Leukemia: a Single Center, Open-label, Controlled Study
Brief Title: Daunorubicin + Cytarabine + Venetoclax in de Novo AML
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Zhangbiao Long, Vice director, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PJ 2023-09-19
Record Dates: First submitted 2024-11-12; First posted 2024-11-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Leukemia, Myeloid, Acute; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Daunorubicin; Cytarabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment(Daunorubicin, Cytarabine, Ventoclax) (Experimental): Treatment(Daunorubicin, Cytarabine, Ventoclax) See Detailed Description.
  Interventions: Drug: (Daunorubicin, Cytarabine, Venetoclax)
- Control(Daunorubicin, Cytarabine) (Active Comparator): Control(Daunorubicin, Cytarabine) See Detailed Description.
  Interventions: Drug: (Daunorubicin, Cytarabine)

INTERVENTIONS:
Drug: (Daunorubicin, Cytarabine, Venetoclax) — * Drugs：Daunorubicin
    * Dosage: 40 mg/(m²·d) on days 1 to 3
    * Other names: Cerubidine, Daunomycin, Rubidomycin
  * Drugs：Cytarabine
    * Dosage: 100 mg/(m²·d) on days 1 to 5
    * Other names: Ara-C, Cytosine Arabinoside, Cytosar-U
  * Drugs：Venetoclax
    * Dosage: 100 mg on day 1, 200 mg on day 2, and 400 mg from days 3 to 14
    * Other names: ABT-199, Venclexta, Venclyxto
  Arms: Treatment(Daunorubicin, Cytarabine, Ventoclax)
Drug: (Daunorubicin, Cytarabine) — * Drugs：Daunorubicin
    * Dosage: 60 mg/(m²·d) on days 1 to 3
    * Other names: Cerubidine, Daunomycin, Rubidomycin
  * Drugs：Cytarabine
    * Dosage: 100 mg/(m²·d) on days 1 to 7
    * Other names: Ara-C, Cytosine Arabinoside, Cytosar-U
  Arms: Control(Daunorubicin, Cytarabine)

SUMMARY:
This study is a non-profit, prospective, single-center, open-label, controlled clinical trial aimed at evaluating the efficacy of the daunorubicin, cytarabine, and venetoclax (DAV) regimen in previously untreated adult AML patients eligible for intensive chemotherapy.The combination of daunorubicin administered for 3 consecutive days and cytarabine for 7 consecutive days constitutes the classic "3+7" induction chemotherapy regimen for AML patients eligible for chemotherapy. The addition of venetoclax to the "3+7" regimen has shown promising efficacy in newly diagnosed AML patients suitable for intensive therapy. However, this approach is associated with increased adverse reactions. Based on current clinical studies, we propose a modified approach involving reduced-dose chemotherapy combined with venetoclax for AML treatment, aiming to achieve optimal efficacy while effectively reducing adverse reactions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1. To evaluate the efficacy of the regimen, as defined by complete remission (CR), complete remission with partial hematologic recovery (CRh), complete remission with incomplete hematologic recovery (CRi), morphological leukemia-free state (MLFS), and partial remission (PR).

SECONDARY OBJECTIVES:

1. To evaluate the long-term effectiveness and durability of the treatment of the regimen, as defined by 1-year overall survival (OS), 1-year event-free survival (EFS), and duration of remission (DOR).
2. To evaluate the safety of the regimen, as defined by Grade 3-4 clinical adverse events (AEs), incidence of laboratory abnormalities, and treatment-related mortality (TRM).

OUTLINE:

* The regimen for the control group includes:(Daunorubicin, Cytarabine)

  * Daunorubicin: 60 mg/(m²·d) on days 1 to 3
  * Cytarabine: 100 mg/(m²·d) on days 1 to 7
* The experimental group's "DAV" regimen includes: (Daunorubicin, Cytarabine, Venetoclax)

  * Daunorubicin: 40 mg/(m²·d) on days 1 to 3
  * Cytarabine: 100 mg/(m²·d) on days 1 to 5
  * Venetoclax: 100 mg on day 1, 200 mg on day 2, and 400 mg from days 3 to 14
* The "DAV" regimen is designed to shorten the duration of induction chemotherapy while extending the application period of venetoclax, aiming to improve efficacy while reducing adverse effects.

ELIGIBILITY:
Inclusion Criteria:(All of the following criteria must be met.)

Patients with newly diagnosed AML based on FAB classification and flow cytometry standards who are eligible for intensive chemotherapy:

* Age between 18 and 59 years;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or 3;
* Expected survival time of ≥3 months;
* None of the following severe cardiac, pulmonary, hepatic, or renal conditions:

  * History of heart disease requiring treatment for congestive heart failure, or an ejection fraction ≤50%, or chronic stable angina;
  * Pulmonary diffusing capacity of carbon monoxide (DLCO) ≤65%, or forced expiratory volume in 1 second (FEV1) ≤65%;
  * Moderate liver impairment with total bilirubin >1.5 to ≤3.0 × the upper limit of normal (ULN);
  * Creatinine clearance ≥30 mL/min to <45 mL/min;
* Has not received radiotherapy, chemotherapy, targeted therapy, or hematopoietic stem cell transplantation within 4 weeks prior to enrollment;
* Has other comorbidities that, in the physician's judgment, make intensive chemotherapy unsuitable;
* Is capable of understanding and willing to sign the informed consent form for this study.

Exclusion Criteria:(Any of the following criteria will exclude the patient from participation)

* Presence of other malignancies;
* Prior treatment with venetoclax or azacitidine;
* History of angioplasty or stent placement within 12 months prior to signing the informed consent, or a history of myocardial infarction, unstable angina, or other clinically significant heart disease;
* Clinically uncontrolled active infection (including bacterial, fungal, or viral infections);
* Pregnant or breastfeeding women;
* Participation in any other clinical trial within 3 months prior to signing the informed consent;
* Any other condition that, in the investigator's judgment, makes the patient unsuitable for participation in this study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | End of cycle 2 (each cycle is 14 days)
  Defined as the proportion of patients achieving complete remission (CR), complete remission with partial hematologic recovery (CRh), complete remission with incomplete hematologic recovery (CRi), morphological leukemia-free state (MLFS), and partial remission (PR) occurring at the end of 2 cycles of treatment. Will be estimated along with the 95% credible interval. Patients who drop out of the study before completing 2 cycles and have been treated will be censored for the primary endpoint analysis.

SECONDARY OUTCOMES:
Overall survival (OS) | 1-Year Follow-up
  Overall survival (OS) is defined as the time from randomization to death from any cause. Patients who are alive at the time of the last follow-up will be censored at the date of last contact. OS will be estimated using Kaplan-Meier methods, with median survival and 95% confidence intervals reported for each treatment group.
Event-free survival (EFS) | 1-Year Follow-up
  Event-Free Survival (EFS) is defined as the time from randomization to the first occurrence of disease progression, relapse, new cancer occurrence, or death from any cause. Patients who remain event-free at the last follow-up will be censored at the date of last contact. EFS will be estimated using Kaplan-Meier methods, with median EFS and 95% confidence intervals reported for each treatment group.
duration of remission (DOR) | 1-Year Follow-up
  Duration of Remission (DOR) is defined as the time from the first documentation of complete or partial remission until disease progression or relapse. Patients who remain in remission at the last follow-up will be censored at the date of last contact. DOR will be estimated using Kaplan-Meier methods, with median DOR and 95% confidence intervals reported for each treatment group.
Incidence of adverse events | 1-Year Follow-up
  Incidence of adverse events will be defined by Grade 3-4 clinical adverse events (AEs), incidence of laboratory abnormalities, and treatment-related mortality (TRM).

CONTACTS AND LOCATIONS:
Overall Officials: ZhangBiao Long, Doctor, Study Chair — Department of Hematology, The First Affiliated Hospital of Anhui Medical University, 218 Jixi Road
Locations (1):
- Department of Hematology, The First Affiliated Hospital of Anhui Medical University, 218 Jixi Road, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
Data Privacy and Ethical Restrictions: The individual participant data collected in this study involves sensitive information. Although de-identification processes have been applied, further measures are required to ensure compliance with relevant ethical standards and data privacy regulations, such as GDPR. We are currently working with ethical committees and relevant authorities to develop a compliant data-sharing strategy.
  Data Quality and Preparation: The data has not yet undergone complete standardization and cleaning processes, and it may not meet the high-quality standards required for sharing. To ensure data accuracy and usability, we plan to consider data sharing once data processing and annotation are fully completed.